CLINICAL TRIAL: NCT01103843
Title: PPD Trial Pilot Study: Plavix, Prasugrel and Drug Eluting Stents
Brief Title: Plavix, Prasugrel and Drug Eluting Stents Pilot Trial
Acronym: PPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Francis Hospital, New York (Other)
Responsible Party: Richard A. Shlofmitz, MD, FACC- Chairman Department of Cardiology, St. Francis Hospital- The Heart Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10-006
Record Dates: First submitted 2010-04-14; First posted 2010-04-15 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2010-04

CONDITIONS: Coronary Artery Disease; Platelet Aggregation Inhibitors; PCI- Percutaneous Coronary Intervention
Keywords: Coronary artery disease; clopidogrel; prasugrel; Verify Now; PRU measurements; Drug eluting stents (EDS); P2Y12; Platelet reactivity
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maintenance Dose Arm (Active Comparator): Open label clopidogrel 75 mg daily or prasugrel 10 mg daily
  Interventions: Drug: Maintenance Dose Arm
- Loading Dose Arm (Active Comparator): Clopidogrel 600 mg or Prasugrel 60 mg at time of PCI.
  Interventions: Drug: Loading Dose Arm

INTERVENTIONS:
Drug: Loading Dose Arm — Subjects who are thienopyridine naive will be randomized 1:1 to either clopidogrel 600 mg or prasugrel 60 mg loading dose at the time of PCI. A Verify Now P2Y12 platelet assay will measure platelet reactivity. Cross over to loading dose and maintenance dose of alternate medication will occur based on level of platelet reactivity.
  Other Names: clopidogrel; prasugrel; Verify now P2Y12 platelet assay
  Arms: Loading Dose Arm
Drug: Maintenance Dose Arm — Verify Now P2Y12 platelet assay will measure platelet reactivity. Cross over to a loading dose and maintenance dose of alternate medication will occur based on level of platelet reactivity.
  Other Names: thienoyridine; Verify now P2Y12; prasugrel; clopidogrel
  Arms: Maintenance Dose Arm

SUMMARY:
* The purpose of this study is to determine the level of inhibition of platelet activation of an approved thienopyridine(clopidogrel or prasugrel) and aspirin regimen in the setting of drug eluting coronary stent implantation.
* In subjects with high residual levels of platelet reactivity after receiving either a maintenance or loading dose of either clopidogrel or prasugrel, a cross over of thienopyridine treatment to the alternate medication will occur.
* The study tests the hypothesis that adequate platelet inhibition will occur in subjects who have high levels of platelet reactivity and are subsequently switched from clopidogrel to prasugrel(loading or maintenance dose) without increased episodes of bleeding or MACE events at discharge and 30 days post Percutaneous Coronary Intervention (PCI).

ELIGIBILITY:
Inclusion Criteria:

* Subject presenting for clinically indicated PCI with implantation of at least one drug-eluting stent.
* No planned use of Glycoprotein IIb/IIIa inhibitors during PCI procedure.
* Subject must be taking aspirin or enteric coated aspirin 81 mg-325 mg daily.
* Willing to participate and sign an informed consent.

Exclusion Criteria:

* Subject older than 75 years of age.
* Subject weight is 60 kg or less.
* Subject who have received intravenous eptifibatide or tirofiban within 48 hours prior to PCI or abciximab within 14 days before or during PCI.
* Subject taking warfarin or with clinical indication to resume warfarin post PCI for any indication.
* Subject currently requiring daily treatment with NSAID or COX2 inhibitors.
* Subject with a known platelet disorder.
* Subject with known active pathological bleeding or heightened risk of bleeding including but not limited to: gastrointestinal bleeding within 6 months, recent surgery or trauma.
* Subject with a history of a stroke or TIA
* Subject with pre-PCI hematocrit or platelet count outside the ranges validated for Verify Now P2Y12 test (33-52% and 119.000-502.000/μL, respectively).
* Subject with a history of hepatic impairment
* Subject with known NYHA Class III or greater for heart failure.
* Inability of subject to provide informed consent.
* Subject with known hypersensitivity or contraindication to clopidogrel, prasugrel or ASA, which would result in inability of patient to adhere to trial protocol.
* Presence of valvular heart disease left main coronary artery stenosis or urgent need for CABG.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-04 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Change in platelet reactivity after switching medication regimen of two thienopyridines- clopidogrel and prasugrel | 4 hours post medicaton administration
  Platelet reactivity will be measured using the Accumetrics Verify Now P2Y12 platelet assay

SECONDARY OUTCOMES:
Occurrence of all bleeding events for subjects enrolled into the trial | 24 hours post PCI or at time of discharge and 30 days post PCI
  All bleeding events will be observed, reported and adjudicated by the DSMB
Occurrence of all MACE events for subjects enrolled into the trial | 24 hours post PCI or at time of discharge and 30 days post PCI
  All bleeding events will be observed, reported and adjudicated by the DSMB

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Shlofmitz, MD, Principal Investigator — Saint Francis Hospital
Locations (1):
- St. Francis Hospital, Roslyn, New York, United States

REFERENCES:
- [Background] Brandt JT, Close SL, Iturria SJ, Payne CD, Farid NA, Ernest CS 2nd, Lachno DR, Salazar D, Winters KJ. Common polymorphisms of CYP2C19 and CYP2C9 affect the pharmacokinetic and pharmacodynamic response to clopidogrel but not prasugrel. J Thromb Haemost. 2007 Dec;5(12):2429-36. doi: 10.1111/j.1538-7836.2007.02775.x. Epub 2007 Sep 26. PMID 17900275
- [Background] Neubauer H, Lask S, Engelhardt A, Mugge A. How to optimise clopidogrel therapy? Reducing the low-response incidence by aggregometry-guided therapy modification. Thromb Haemost. 2008 Feb;99(2):357-62. doi: 10.1160/TH07-10-0624. PMID 18278186
- [Background] Gurbel PA, Bliden KP, Hiatt BL, O'Connor CM. Clopidogrel for coronary stenting: response variability, drug resistance, and the effect of pretreatment platelet reactivity. Circulation. 2003 Jun 17;107(23):2908-13. doi: 10.1161/01.CIR.0000072771.11429.83. Epub 2003 Jun 9. PMID 12796140
- [Background] Ferguson AD, Dokainish H, Lakkis N. Aspirin and clopidogrel response variability: review of the published literature. Tex Heart Inst J. 2008;35(3):313-20. PMID 18941611
- [Background] Simon T, Verstuyft C, Mary-Krause M, Quteineh L, Drouet E, Meneveau N, Steg PG, Ferrieres J, Danchin N, Becquemont L; French Registry of Acute ST-Elevation and Non-ST-Elevation Myocardial Infarction (FAST-MI) Investigators. Genetic determinants of response to clopidogrel and cardiovascular events. N Engl J Med. 2009 Jan 22;360(4):363-75. doi: 10.1056/NEJMoa0808227. Epub 2008 Dec 22. PMID 19106083
- [Background] Farid NA, Kurihara A, Wrighton SA. Metabolism and disposition of the thienopyridine antiplatelet drugs ticlopidine, clopidogrel, and prasugrel in humans. J Clin Pharmacol. 2010 Feb;50(2):126-42. doi: 10.1177/0091270009343005. Epub 2009 Nov 30. PMID 19948947
- [Background] Wiviott SD, Braunwald E, McCabe CH, Montalescot G, Ruzyllo W, Gottlieb S, Neumann FJ, Ardissino D, De Servi S, Murphy SA, Riesmeyer J, Weerakkody G, Gibson CM, Antman EM; TRITON-TIMI 38 Investigators. Prasugrel versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2007 Nov 15;357(20):2001-15. doi: 10.1056/NEJMoa0706482. Epub 2007 Nov 4. PMID 17982182
- [Background] Wiviott SD, Trenk D, Frelinger AL, O'Donoghue M, Neumann FJ, Michelson AD, Angiolillo DJ, Hod H, Montalescot G, Miller DL, Jakubowski JA, Cairns R, Murphy SA, McCabe CH, Antman EM, Braunwald E; PRINCIPLE-TIMI 44 Investigators. Prasugrel compared with high loading- and maintenance-dose clopidogrel in patients with planned percutaneous coronary intervention: the Prasugrel in Comparison to Clopidogrel for Inhibition of Platelet Activation and Aggregation-Thrombolysis in Myocardial Infarction 44 trial. Circulation. 2007 Dec 18;116(25):2923-32. doi: 10.1161/CIRCULATIONAHA.107.740324. Epub 2007 Dec 3. PMID 18056526
- [Background] Li YG, Ni L, Brandt JT, Small DS, Payne CD, Ernest CS 2nd, Rohatagi S, Farid NA, Jakubowski JA, Winters KJ. Inhibition of platelet aggregation with prasugrel and clopidogrel: an integrated analysis in 846 subjects. Platelets. 2009 Aug;20(5):316-27. doi: 10.1080/09537100903046317. PMID 19637095
- [Background] Mega JL, Close SL, Wiviott SD, Shen L, Hockett RD, Brandt JT, Walker JR, Antman EM, Macias WL, Braunwald E, Sabatine MS. Cytochrome P450 genetic polymorphisms and the response to prasugrel: relationship to pharmacokinetic, pharmacodynamic, and clinical outcomes. Circulation. 2009 May 19;119(19):2553-60. doi: 10.1161/CIRCULATIONAHA.109.851949. Epub 2009 May 4. PMID 19414633
- [Background] Payne CD, Li YG, Brandt JT, Jakubowski JA, Small DS, Farid NA, Salazar DE, Winters KJ. Switching directly to prasugrel from clopidogrel results in greater inhibition of platelet aggregation in aspirin-treated subjects. Platelets. 2008 Jun;19(4):275-81. doi: 10.1080/09537100801891640. PMID 18569863
- [Background] Godino C, Mendolicchio L, Figini F, Latib A, Sharp AS, Cosgrave J, Calori G, Cera M, Chieffo A, Castelli A, Maseri A, Ruggeri ZM, Colombo A. Comparison of VerifyNow-P2Y12 test and Flow Cytometry for monitoring individual platelet response to clopidogrel. What is the cut-off value for identifying patients who are low responders to clopidogrel therapy? Thromb J. 2009 May 6;7:4. doi: 10.1186/1477-9560-7-4. PMID 19419580